CLINICAL TRIAL: NCT06560957
Title: Feasibility and Acceptability of Adjunctive Time Restricted Eating in Bipolar Disorder: a Pilot Randomized Controlled Trial.
Brief Title: SYNCED - SYNChronized Eating in Bipolar Depression Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Gayatri Saraf, Psychiatrist and Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240310-01H
Record Dates: First submitted 2024-06-12; First posted 2024-08-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Eating ad libitum, nutritional counselling plus treatment as usual (Other): Participants randomized to this group will be offered nutritional counselling from a registered dietician. They will also receive a check-in from the registered dietician at week 4. They will also continue to receive treatment as usual. Treatment as usual includes pharmacological treatment options such as mood stabilizers and/or atypical antipsychotics, and psychological treatments such as psychotherapy. No current treatments will be stopped to participate in the study. We will record changes made to the doses of medications during the trial. No new treatments will be started for the duration of the trial, including pharmacological and psychological treatments
  Interventions: Behavioral: Eating ad libitum with nutritional counselling
- Group 2:Time-restricted eating plus treatment as usual (Other): In addition to the nutritional counselling and continuing treatment as usual outlined in Group 1, this group will be provided time restricted eating instruction. The experimental group will be instructed to select a consistent 10-h eating window between 06:00 and 19:00 for all days of the week to consume all food and beverages (except water) for the duration of the 8-week intervention. Adherence to the intervention will be monitored weekly through phone check-ins with the research assistant. At 4-weeks, the study dietician will have a 1-hour check in with participants to review progress and adherence to TRE and to address any difficulties the participants may be facing.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Time restricted eating involves restricting the window in which calories are consumed to 8-10 hours, without altering diet quality or caloric intake. In this study, time restricted eating will be a consistent 10-h eating window between 06:00 and 19:00, considered an early TRE pattern, for all days of the week, as chosen by the participant. They will need to consume all food and beverages (except water) during this window for the duration of the 8-week intervention.
  Arms: Group 2:Time-restricted eating plus treatment as usual
Behavioral: Eating ad libitum with nutritional counselling — Nutritional counselling will include customized advice delivered by a registered dietician about dietary choices while allowing individuals to eat at any time of day.
  Arms: Group 1: Eating ad libitum, nutritional counselling plus treatment as usual

SUMMARY:
Bipolar disorders (BD) are a group of complex disorders that impact mood, behaviour and cognition and are known to cause significant suffering and impairment. Circadian rhythm (your internal day/night "clock") disruption, which can involve changes in sleep-wake cycles, frequently occurs in BD. Both depression and mania are accompanied by circadian disruption. These disruptions are hypothesized to lead to mood worsening, metabolic dysfunction and inflammation. If circadian dysfunction plays a significant role in the symptoms and trajectory of BD, then treatment approaches that target these functions may lead to better outcomes. One such approach is dietary interventions. Time restricted eating (TRE) is a dietary tool that restricts the eating to an 8-12 hour window, without changing diet quality or caloric intake. Studies involving time restricted eating have been done in other conditions with promising results. There have been no studies done for mood disorders in general or bipolar disorder specifically. In this proposal, the investigators will assess two dietary interventions (TRE and nutritional counselling) to examine how TRE may represent a safe and viable adjunct to traditional treatments. The investigators aim to compare TRE with nutritional counselling, while all participants continue to receive usual care. Participants will receive support from a registered dietician and will be instructed on dietary habits. Half of participants will receive nutritional counselling and half will be asked to do TRE. Those in the TRE group will be asked to select a 10-hour window to consume all food and non-water beverages for the 8-week period. Participants will be asked to complete a screening visit to determine eligibility, and then will complete questionnaires at baseline, week 4 and week 8 examining symptoms of their illness and cognition. Participants will also provide a blood sample at baseline and week 8 for standard biochemistry tests, pregnancy testing (if applicable), and to examine inflammatory markers. Participants will also wear an actigraphy watch which provides wireless continuous monitoring of movements and ambient light. The primary outcome is feasibility and acceptability (do people agree to participate, complete the study, and follow the intervention; what do they think of the intervention). Secondary outcomes include changes in depression, anxiety, sleep, and cognition. Exploratory outcomes include inflammatory markers and circadian disruption.

DETAILED DESCRIPTION:
Given the lack of studies evaluating time restricted eating (TRE), this pilot study aims to examine the feasibility and acceptability of TRE as a prelude to a future multi-centre randomized controlled trial (RCT) evaluating efficacy. If adjunctive TRE is found to be feasible, this will pave the way for a novel and safe intervention which may have the potential to treat circadian dysfunction, metabolic side effects and improve mood and cognitive outcomes in patients with BD.

To evaluate the feasibility and acceptability of adjunctive 10-hour TRE with treatment as usual relative to nutritional counselling and treatment as usual for the treatment of depression associated with bipolar disorder. To do this, the investigators will estimate the rate (proportion) of eligible people who are willing to participate, participants who drop out of the trial and participants who adhere to their allocated intervention.

First, the investigators hypothesize that the investigators would achieve our recruitment target of 40 patients with BD within the study's 18-month duration and retain at least 70% of participants through the follow-up period to evaluate feasibility. The investigators will also be able to estimate what level of adherence could be expected following a single intervention with a 4-week reminder. Second, the investigators hypothesize that participants would complete the intervention and find it acceptable.

Secondary Objectives To assess if TRE leads to meaningful reductions in markers of depression, anxiety, sleep, quality of life, and cognition.

The investigators hypothesize a greater reduction in depressive symptoms, anxiety symptoms compared to that seen in the control group. The investigators also hypothesize improvements in sleep, quality of life and cognition compared to the control group.

Exploratory Objectives Effects on inflammatory markers and circadian disruption will be additionally explored.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-55 years old
2. Have a diagnosis of bipolar I or bipolar II disorder, confirmed by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) Research Version (SCID-RV)
3. Have mild to moderate depression symptoms as indicated by a score of ≥12 and ≤30 on MADRS and ≤12 on Young Mania Rating Scale (YMRS).
4. Be willing to use email for study activities
5. Females of childbearing potential are willing to follow highly effective methods of contraception (mentioned below) for the duration of study*
6. Be able and willing to use email and a smartphone application for the duration of the trial
7. Participants must be able to speak, read, write and understand English or French.
8. Be willing and able to provide informed consent.

Exclusion Criteria:

1. Have clinically significant suicidal ideation, defined as ≥ 4 on MADRS suicide item
2. Have any catatonic symptoms, eating disorders, borderline personality disorder and substance use disorders as measured by the Structured Clinical Interview for the DSM-5 Research Version (SCID-RV)
3. Have any unstable or inadequately treated neurological and medical conditions
4. Have had prior bariatric surgery
5. Be taking hypoglycemia inducing medications
6. Be pregnant or lactating
7. Currently on stimulant medications
8. Be participating in any other diet or weight management program for the duration of the trial.
9. Have any contraindication to fasting as judged by the assessing clinician.
10. Recently started taking a Canadian Network for Mood and Anxiety Treatments (CANMAT) recommended treatment18 for the management of acute bipolar depressive episode, but has not had a trial for a minimum of 6 weeks with adequate doses.
11. Recently (i.e. within the past 8 weeks) began structured psychotherapy (i.e. cognitive-behavioral therapy, interpersonal psychotherapy, family-focused therapy, or interpersonal and social rhythm therapy).
12. Have any other medical condition for which physician or investigator team expresses concern about safety or ability to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the study | 18 months
  The investigators will consider the intervention feasible if 70% of participants complete follow-up.
Time to recruit all participants | 18 months
  The investigators will consider the intervention feasible if 70% of participants complete follow-up.
Intervention adherence | 18 months
  The investigators will consider the intervention acceptable if participant adherence to the intervention is at least 70% (i.e. participants adhere to the TRE intervention 40 days out of 56 days); ii) at least 50% of participants approached about the study agree to participate.
Rate of participation | 18 months
  The investigators will consider the intervention acceptable if at least 50% of potential participants approached about the study agree to participate.

SECONDARY OUTCOMES:
Depression severity - Montgomery-Åsberg Depression Rating Scale | Screening, Baseline (week 1), Week 4, Week 8
  The Montgomery-Åsberg Depression Rating Scale (Structured Interview Guide) (MADRS) is a 10-item observer-rated scale to assess the severity of depressive symptoms within the last 7 days. Possible total score range is 0-60. Score of: 0-8 indicates remission/absent symptoms; 9-17 mild depression, 18-34 moderate depression; and 35-60 severe depression.
Cognitive dysfunction - Cognitive Complaints in Bipolar Disorder Rating Assessment | Baseline (week 1), Week 4, Week 8
  A 16-item self-report that assess subjective cognitive dysfunction (including executive function, processing speed, working memory, verbal learning and memory, attention/concentration and mental tracking) in bipolar disorder. Measured on a 4-point Likert scale ranging from never (0) to always (3). Scores range 0-48 with higher scores indicating worse cognitive dysfunction.
Cognitive Dysfunction - Screen for Cognitive Impairment in Psychiatry | Baseline (week 1), Week 4, Week 8
  The Screen for Cognitive Impairment in Psychiatry (SCIP) is a brief clinician administered evaluation of cognitive deficits including working memory, immediate and delayed verbal list learning, verbal fluency, and psychomotor speed. Score is calculated as a sum of 5 subgroups, with subgroup 3 having no limit to the total score. Total score ranges from 0 with no upper limit, with lower scores showing more cognitive impairment. These scores are interpreted in the following manner: total score of < 75 suggest mild impairment, score of < 65 indicate moderate impairment, and score of < 55 indicate severe impairment.
Anxiety severity - Hamilton Anxiety Rating Scale | Baseline (week 1), Week 4, Week 8
  The Hamilton Anxiety Rating Scale (HAM-A) is a 14-item semi-structured observer-rated interview evaluating symptoms of anxiety. Each item is scored 0 (not present) to - 4 (very severe). Scores range 0-56 with higher scoring indicating worse severity of anxiety symptoms. These scores are interpreted in the following manner: scores of 0-7 indicate remission/symptom absence, 8-14 mild anxiety, 15-23 moderate anxiety and 24-56 severe anxiety.
Anxiety severity - Generalized Anxiety Disorder-7 | Baseline (week 1), Week 4, Week 8
  Self-reported measurement of the severity of anxiety symptoms experienced within the last two weeks. It consists of 7 scored items and one follow-up question. Each of the 7 scored items generates a value from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0 to 21, with higher scores indicating more severe symptoms of anxiety. These scores are interpreted in the following manner: a score of 0-4 indicates little or no anxiety, a score of 5-9 indicates mild anxiety, a score of 10-14 indicates moderate anxiety, and a score of 15-21 indicates severe anxiety. Generally, a score of 10 or above is considered to be a clinical cutoff implying that the respondent may be suffering from a general anxiety disorder.
Biological Rhythms - Biological Rhythm Interview for Assessment in Neuropsychiatry | Baseline (week 1), Week 4, Week 8
  A 21-item observer-rated measure that assess five areas related to biological rhythms (sleep, activity, social aspect, diet, and predominant rhythm (chronotype)). All items are evaluated on a 4-point likert scale ranging from 1-4, with higher scores indicating greater disturbance. Total score ranges from 21-84.
Sleep Quality - Reduced Pittsburgh Sleep Quality Index | Baseline (week 1), Week 4, Week 8
  The Pittsburgh Sleep Quality Index Questionnaire is self-administered questionnaire designed to evaluate sleep quality consisting of 18 items that in turn are comprised of seven components, which include subjective sleep quality, sleep duration, sleep onset, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. Each weighted equally on a 0-3 scale to be summed to yield a global PSQI score, which ranges between 0 and 21, where the higher the scores, the worse the sleep quality. The investigators will only be using questions 1-4 and 6 (reduced PSQI).
19-Item Self-Assessment Questionnaire for Sleep Rhythms, Habits and Fatigue (MEQ) | Baseline (week 1), Week 4, Week 8
  This questionnaire has 19 questions, each with a number of points. Scores can range from 16-86. Scores of 41 and below indicate "evening types." Scores of 59 and above indicate "morning types." Scores between 42-58 indicate "intermediate types."
Function - Global Assessment of Functioning | Baseline (week 1), Week 4, Week 8
  A numeric ranking between 0 and 100 that summarizes the clinician's view of the patient's current degree of impairment in terms of psychosocial and occupational or educational function. Higher scores indicate better functioning. Normal functioning typically ranges from 70-100.
Symptom Severity and Improvement - Clinical Global Impressions-BP-Severity & Improvement (CGI-BP I&S) | Baseline (week 1), Week 4, Week 8
  The CGI-BP I&S is a measure of CGI-I and CGI-S specifically validated for bipolar disorder. The CGI-BP-S scale provides a brief assessment of the severity of a patient's mental illness at baseline and following treatment. CGI-I and CGI-S are each rated on a likert scale of 0-7 (0, not assessed, 1-7 normal to most extremely ill). The CGI-BP-I scale provides a brief assessment of a patient's overall mental state following treatment, and whether or not it is due entirely to the experimental treatment.
Psychological Dysfunction - Functioning assessment short test (FAST) | Baseline (week 1), Week 4, Week 8
  The FAST is a brief clinician-reported scale which assess psychosocial dysfunction across multiple domains (autonomy, occupational functioning, cognitive functioning, financials, interpersonal relationships, and leisure time) in people with bipolar disorder. Aspects of functioning are rated on a 4-point Likert scale of 0 (no difficulty) to 3 (severe difficulty) with total scores ranging from 0-72. Higher scores indicate more dysfunction.
Quality of Life - Brief Quality of Life in Bipolar Disorder Questionnaire | Baseline (week 1), Week 4, Week 8
  A brief 12-item self report that examines quality of life in people living with bipolar disorder over the past 7 days. Experiences of quality of life are rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly Agree). Total scores range from 12-60 with higher scores indicating better quality of life.
Mania severity - Young Mania Rating Scale | Screening, Baseline (week 1), Week 4, Week 8
  The Young Mania Rating Scale is used to evaluate the severity of manic symptoms at baseline and over time in individuals with mania. It is an 11-item scale and total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).

OTHER OUTCOMES:
Change in circadian rhythms | Week 0, Week 9
  Using wrist actigraphy, the investigators will collect data on two 24-hour sleep-wake cycles. The validated wrist actigraphy monitor will collect non-invasive, wireless continuous monitoring of movements and ambient light (in the blue, green and red spectrum). These two measures will be combined to extract sleep estimates and parameters of the 24-hour activity-rest cycle before and after the intervention. Changes in the circadian rhythms (hours of sleep or movement) will be compared pre- and post between treatment groups.
Change in C-reactive protein levels | Baseline (week 1), Week 8
  The investigators will collect blood samples and measure levels of C-reactive protein (CRP) before and after the intervention. CRP is an inflammation marker and measured in mg/L.
Change in cytokine levels | Baseline (week 1), Week 8
  The investigators may collect blood samples and measure levels of cytokines including interleukins (IL) -6, IL-10, IL-1B and tumor necrosis factor alpha (TNF-a) before and after the intervention. IL-6, IL-10 and TNF-a are inflammatory cytokines and IL-10 is an anti-inflammation cytokine. All cytokines are measured in pg/mL.
Change in red blood cell count | Baseline (week 1), Week 8
  The investigators will collect blood samples to evaluate changes in red blood cell count (RBC) as part of changes in hematology before and after intervention. This will be done as part of a complete blood count (CBC) will be conducted to investigate changes in various blood components. RBC is measured in x10*12/L
Change in hemoglobin | Baseline (week 1), Week 8
  The investigators will collect blood samples to evaluate changes in hemoglobin (Hgb) as part of changes in hematology before and after intervention. This will be done as part of a complete blood count (CBC) will be conducted to investigate changes in various blood components. Hgb is measured in g/L.
Change in hematocrit | Baseline (week 1), Week 8
  The investigators will collect blood samples to evaluate changes in hematocrit (Hct) as part of changes in hematology before and after intervention. This will be done as part of a complete blood count (CBC) will be conducted to investigate changes in various blood components. Hct is measured in L/L..
Change in lymphocyte count | Baseline (week 1), Week 8
  The investigators will collect blood samples to evaluate changes in lymphocyte count as part of changes in hematology before and after intervention. This will be done as part of a complete blood count (CBC) will be conducted to investigate changes in various blood components. Lymphocyte count is measured in x10*9/L.
Change in blood chemistry | Baseline (week 1), Week 8
  The investigators may collect blood samples to evaluate changes in blood chemistry before and after the intervention. The test will include fasting glucose, fasting lipid profile (includes measures of high-density and low-density lipoprotein cholesterol, total cholesterol and triglycerides). All blood chemistry measures are measured in mmol/L.
Change in liver functions | Baseline (week 1), Week 8
  The investigators may collect blood samples to evaluate changes in liver function by measuring alkaline phosphatase (ALP), aspartate transferase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT) before and after the intervention. All measures are reported in U/L.
Change in total bilirubin | Baseline (week 1), Week 8
  The investigators may collect blood samples to evaluate changes in liver function by measuring total bilirubin before and after the intervention. This is measured in umol/L.
Change in serum creatinine | Baseline (week 1), Week 8
  The investigators will collect blood samples to evaluate changes in blood chemistry by measuring total serum creatinine before and after the intervention. This is measured in umol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Gayatri Saraf, MD, Principal Investigator — The Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No